CLINICAL TRIAL: NCT04674969
Title: Drug-Eluting Registry: Real-World Treatment of Lesions in the Peripheral Vasculature (ELEGANCE)
Brief Title: Drug-Eluting Registry: Real-World Treatment of Lesions in the Peripheral Vasculature
Acronym: ELEGANCE
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2444
Record Dates: First submitted 2020-12-01; First posted 2020-12-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Clinical Cohort: All enrolled patients are included in the Clinical Cohort. Patients will complete assessments per standard of care through 2-year follow-up in Australia, Austria, Canada, France, Germany, Poland, Spain, Taiwan, Thailand, and the United States. Patients will complete assessments per standard of care through 5-year follow-up in China.
  Interventions: Device: Any eligible commercially available Boston Scientific Corporation (BSC) drug-eluting device.
- Outcomes Cohort: Patients at select sites will complete the Clinical Cohort standard of care assessments and additional assessments as part of the Outcomes Cohort, including Quality of Life questionnaires, six-minute walk test (6MWT), and Healthcare Utilization data collection.
  Interventions: Device: Any eligible commercially available Boston Scientific Corporation (BSC) drug-eluting device.

INTERVENTIONS:
Device: Any eligible commercially available Boston Scientific Corporation (BSC) drug-eluting device. — Ranger™ Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter; ELUVIA™ Drug-Eluting Vascular Stent System

SUMMARY:
The ELEGANCE Registry's objective is to collect Real-World Data (RWD), including populations previously not represented in Peripheral Vascular Disease (PVD) trials, health economics data, and to support the safe use of commercially available Boston Scientific Corporation (BSC) drug-eluting devices for the treatment of lesions located in the peripheral vasculature.

DETAILED DESCRIPTION:
A global prospective, non-randomized, open-label, multi-center Registry to collect Real-World Data, including health economic data, to support the use of commercially available drug-eluting BSC devices for the treatment of lesions located in the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Written informed consent (patient data release-form)
* Use of any commercially available Boston Scientific drug-eluting device marketed for treatment of lesions in the peripheral vasculature and specified in the Registry Enrollment Guide

Exclusion Criteria:

* Life expectancy of <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population for the ELEGANCE Registry are real-world patients who are treated with commercially available BSC drug-eluting devices marketed for treatment of lesions located in the peripheral vasculature. Efforts will be made to include study centers with diverse patient populations in order to enroll populations previously not represented in PVD trials.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | 12 months
  Rate of MAEs, which include Target Lesion Revascularizations, Major Target Limb Amputations, and Deaths. No pre-specified endpoints or formal tests of hypotheses are proposed. Analyses will be performed for exploratory purposes.
Lesion Patency | 12 months
  Lesion patency is determined by Duplex Ultrasound (Investigator and/or Core Lab assessed) and freedom from clinically-driven Target Lesion Revascularization. No pre-specified endpoints or formal tests of hypotheses are proposed. Analyses will be performed for exploratory purposes.

CONTACTS AND LOCATIONS:
Locations (79):
- United States (52):
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - PIH Health Good Samaritan Hospital, Los Angeles, California
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - Adventist Health St Helena Hospital, St. Helena, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newport, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Heart & Vascular, LLC, Boynton Beach, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Rush University, Chicago, Illinois
  - St. John's Hospital/ Prairie Education and Research Cooperative, Springfield, Illinois
  - St. Joseph Hospital/Dupont Hospital, Fort Wayne, Indiana
  - Ascension St. Vincent's Hospital, Indianapolis, Indiana
  - CIS Clinical Research Corporation, Houma, Louisiana
  - Ochsner Clinic Foundation, Kenner, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mercy Hospital (Allina Health), Coon Rapids, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Buffalo General Hospital, Buffalo, New York
  - North Shore University Hospital/Northwell Health, Manhasset, New York
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Hospital, New York, New York
  - Weill Cornell Medicine/New York-Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rex UNC Health (NC Heart and Vascular Research, LLC), Raleigh, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Premier Cardiovascular Institute, Dayton, Ohio
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Hospital University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota
  - Seton Medical Center, Austin, Texas
  - The University of Texas, Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - HeartPlace P.A., Plano, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
  - UW Medicine - Harborview Medical Center, Seattle, Washington
- Australia (2):
  - Royal Perth Hospital, Perth, Western Australia
  - Royal North Shore Hospital, St Leonards
- Medizinische Univ.-Kliniken Graz, Graz, Austria
- Canada (2):
  - Peter Lougheed Centre-Hospital, Calgary, Alberta
  - CHUS - Hotel Dieu, Sherbrooke, Quebec
- China (11):
  - Beijing Anzhen Hospital of the Capital University of Medical Sciences, Chaoyang, Beijing Municipality
  - China-Japan Friendship Hospital, Chaoyang, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Xicheng, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan University No.1 Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - Shanghai Ninth People's Hospital - Shanghai Jiaotong University School of Medicine, Huangpu, Shanghai Municipality
  - Shanghai Changhai Hospital, Yangpu, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanghai Zhongshan Hospital, Shanghai, Xuhui District
- France (2):
  - Hospital Marie Lannelongue, Le Plessis-Robinson
  - Hospital Paris Saint Joseph, Paris
- Germany (3):
  - Fürst Stirum Klinik Bruchsal Hospital, Bruchsal
  - University Clinic Essen-Hospital, Essen
  - Klinikum der Ludwig-Maximilians-Universitat, München
- Uniwersyteckim Szpitalem Klinicznym w Poznaniu, Poznan, Poland
- Corporacio Sanitaria Parc Taulí, Barcelona, Sabadell, Spain
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Siriraj Hospital Department of Surgery, Bangkok
  - Prince of Songkla University, Hat Yai

REFERENCES:
- [Derived] Secemsky EA, Giri J, Brodmann M, Goueffic Y, Fu W, Greenberg-Worisek AJ, Jaff MR, Kirksey L, Kohi MP. Implementing methods in the ELEGANCE registry to increase diversity in clinical research. J Vasc Surg. 2024 Jan;79(1):136-145.e3. doi: 10.1016/j.jvs.2023.08.131. Epub 2023 Sep 22. PMID 37742734